CLINICAL TRIAL: NCT06143241
Title: The Effect of Respiratory Muscle Performance on Cognitive Functions in Children with Epilepsy: Monitoring with Glymphatic System Activation and Neuropeptides
Brief Title: Cognitive Function and Glymphatic System in Children with Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Miray Baser, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16.11.2023
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy; Cognitive Dysfunction; Seizure, Epileptic
Keywords: Cognition; Epilepsy; Glymphatic System; Breathing Exercises
MeSH Terms: conditions — Epilepsy; Cognitive Dysfunction; Seizures

STUDY DESIGN:
Intervention Model Description: Children diagnosed with epilepsy will be divided into two groups as experimental group and control group using block randomisation method.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be informed about the intergroup practice. The person who will carry out the evaluations will not be informed about the application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): It consists of 20 children diagnosed with epilepsy who will receive inspiratory muscle training following routine medication use. The experimental group will receive inspiratory muscle training with the Thershold device for 30 minutes every day for 8 weeks.
  Interventions: Device: Threshold IMT; Drug: Antiepileptic medication
- Control Group (Active Comparator): The control group consists of 20 children diagnosed with epilepsy who will only be followed up with routine medication.
  Interventions: Drug: Antiepileptic medication

INTERVENTIONS:
Device: Threshold IMT — Threshold is used in respiratory muscle training in the form of resistance loading.
  Arms: Experimental Group
Drug: Antiepileptic medication — They will continue their antiepileptic medication prescribed by their doctor.

SUMMARY:
Epilepsy, one of the most common neurological disorders in childhood, is a chronic brain disease characterized by neurobiological, psychological and cognitive effects. Neuropeptide-Y (NPY) and neural growth factor (NGF) play a role in different pathological processes seen in epileptogenesis. Neuron-specific enolase (NSE), a quantitative indicator of brain damage, has been shown to exhibit elevated serum levels in individuals with epilepsy and is associated with cognitive functions.

It is reported that the glymphatic system, which is associated with epileptic seizures, is a treatment method that can prevent cognitive impairment by preventing the accumulation of toxic waste proteins.

Inspiratory muscle training, one of the respiratory physiotherapy techniques, is used as supportive treatment in patients with weak respiratory muscle strength. Weakness in respiratory muscle strength has also been detected in the epilepsy group in which the glymphatic system is affected.

40 children with epilepsy who meet the inclusion criteria and volunteer to participate in the study will participate. Children with epilepsy will be divided into two groups: experimental group (n = 20) and control group (n = 20) using the block randomization method.

The experimental group will be given Inspiratory Muscle Training (IMT) with the Threshold device for 30 minutes every day for 8 weeks after routine medication use. The control group will be followed only with routine medication use.

Demographic information of all participants will be recorded. Respiratory function will be evaluated with a portable spirometer device, respiratory muscle strength will be evaluated with a portable electronic mouth pressure measurement device, and cognitive performance will be evaluated with the Serial Digit Learning Test (SDLT).

Biochemical analyses; Serum levels of neuron specific enolase (NSE), neuropeptide-Y (NPY) and neural growth factor (NGF) will be determined with an ELISA kit set. The glymphatic system will be evaluated with Diffusion Tensor Imaging Analysis Across the Perivascular Space (DTI-ALPS). In both groups, the initial evaluations will be repeated after 8 weeks.

This research project was planned to prevent the development of seizures and improve biochemical parameters, glymphatic system dysfunction and cognitive functions with inspiratory muscle training in pediatric epilepsy patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with absence and rolandic type epilepsy according to the International League Against Epilepsy (ILAE) classification.
* No previous respiratory physiotherapy.
* Maximal Inspiratory Pressure (MIP) value is below the expected value according to age and gender.
* Co-operative.

Exclusion Criteria:

* Diagnosed with respiratory system disease.
* Has kyphoscoliosis and/or advanced postural alignment problems that affect respiratory function.
* Have severe mental problems.
* Receiving ketogenic diet application.
* Have any neuromuscular disease.
* Have severe cardiac involvement, pulmonary embolism, mesenteric or portal thrombosis.
* Diagnosis of inflammatory disease or C-reactive protein (CRP) analysis above normal limits.
* The presence of orthopedic surgery.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  Respiratory muscle strength will be measured according to American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria using a portable electronic mouth pressure measurement device (micro RPM). A measurement result of 80 cmH2O and above indicates a good result.
Spirometer | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  It will be performed using a portable spirometer (Cosmed Pony FX, Italy). The test will be performed in a seated position with the patient being asked to first take a deep breath and then exhale rapidly into the spirometer device. A nose clip will be used during exhalation. The forced vital capacity (FVC) value will be recorded in litres and %.
Spirometer | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  It will be performed using a portable spirometer (Cosmed Pony FX, Italy). The test will be performed in a seated position with the patient being asked to first take a deep breath and then exhale rapidly into the spirometer device. A nose clip will be used during the exhalation. The forced expiratory volume in one second (FEV1) value will be recorded in litres and %.
Spirometer | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  It will be performed using a portable spirometer (Cosmed Pony FX, Italy). The test will be performed in a seated position with the patient being asked to first take a deep breath and then exhale rapidly into the spirometer device. A nose clip will be used during the exhalation. The forced expiratory volume in one second/forced vital capacity (FEV1/FVC) value will be recorded in litres and %.
Spirometer | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  It will be performed using a portable spirometer (Cosmed Pony FX, Italy). The test will be performed in a seated position with the patient being asked to first take a deep breath and then exhale rapidly into the spirometer device. A nose clip will be used during exhalation. The peak expiratory flow (PEF) value will be recorded in litres and %.
Neuron specific enolase (NSE) | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  Blood samples will be collected interictal and serum will be separated and stored. Analyses will be performed by ELISA.
Neuropeptide-Y (NPY) | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  Blood samples will be collected interictal and serum will be separated and stored. Analyses will be performed by ELISA.
Neural growth factor (NGF) | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  Blood samples will be collected interictal and serum will be separated and stored. Analyses will be performed by ELISA.
Serial Digit Learning Test (SDLT) | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  Evaluates short-term memory and learning ability. In the test content, there are two separate sequences of 8 or 9 digits in which the digits from 1 to 9 are mixed according to the age and education level of the participant. The selected sequence is read to the subject in order and the subject is asked to remember and say the sequence in the correct order.
Diffusion Tensor Imaging Analysis Across Perivascular Space (DTI-ALPS) | It will be measured at baseline and at the end of the experiment (at the end of 8 weeks).
  It is used to measure glymphatic system activation. A rectangular ROI is drawn and fiber orientations and diffusivities in all three directions along the x-, y-, and z-axes are obtained as voxel levels. Among several voxels, for each fiber on the same x-axis (projection, association, and subcortical fibers), one voxel is selected that shows the most common orientation in each fiber. The DTI-ALPS index is the average of two sets of diffusivity values perpendicular to the dominant fibers in the tissue, namely the x-axis diffusivity in the area of projection fibers (Dxproj) and the x-axis diffusivity in the area of association fibers (Dxassoc), the y-axis diffusivity in the area of projection fibers (Dyproj) and the area of association fibers. It is calculated as the ratio of the z-axis diffusivity (Dzaccoc) to its average.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
At the end of the research, the data of the participants and the details of the protocol applied can be requested from the responsible researcher via e-mail address in line with the necessary justifications.
Supporting Information: Study Protocol